CLINICAL TRIAL: NCT06635967
Title: The Efficacy of Repetitive Transcranial Magnetic Stimulation in Patients With Chronic Subjective Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024098
Record Dates: First submitted 2024-10-09; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-08

CONDITIONS: Tinnitus
Keywords: tinnitus; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- frequency-specific patterned rTMS (Experimental): Patients will receive a 5-day, once-daily frequency-specific patterned rTMS treatment via a circular coil applied to the auditory cortex. Each session will last 40 minutes and will be stimulated at an intensity of 80% resting motor threshold (RMT).
  Interventions: Device: frequency-specific rTMS
- 1 Hz rTMS (Active Comparator): Patients will receive a 5-day, once-daily 1Hz rTMS treatment via a circular coil applied to the auditory cortex. Each session will last 40 minutes and will be stimulated at an intensity of 80% resting motor threshold (RMT).
  Interventions: Device: 1 Hz rTMS

INTERVENTIONS:
Device: frequency-specific rTMS — Patterned repetitive transcranial magnetic stimulation will be performed at specific frequencies and inter-train intervals
  Arms: frequency-specific patterned rTMS
Device: 1 Hz rTMS — Low-frequency rTMS will be performed at a frequency of 1Hz
  Arms: 1 Hz rTMS

SUMMARY:
The aim of this study is to compare the efficacy of frequency-specific patterned repetitive transcranial magnetic stimulation (rTMS) and 1Hz rTMS for the treatment of chronic subjective tinnitus. In this single-blind randomized controlled study, patients will be randomly assigned 1:1 to receive two different types of rTMS stimulation.

DETAILED DESCRIPTION:
Tinnitus is a common disorder with a prevalence of 10-25% among adults, which seriously affects the quality of life of patients. Many studies have reported significant efficacy of repetitive transcranial magnetic stimulation (rTMS) for tinnitus, but its optimal stimulation parameters are not clear. Therefore, there is necessary to assess the clinical efficacy and mechanism of different types of rTMS for the treatment of chronic subjective tinnitus through rigorously designed clinical studies.

The study will assess the severity of tinnitus and the mood and sleep status of the patients through several scales and tinnitus psychoacoustic assessment before treatment, after treatment and at follow-up. The primary research hypothesis is that frequency-specific patterned rTMS will be superior to 1Hz rTMS in reducing tinnitus-related distress.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 80 years old.
2. Experiencing persistant subjective tinnitus for at least 3 months.
3. A score of 38 or more on THI.
4. 50 dB HL or less on the average pure tone threshold (0.5, 1, 2kHz) of the worse ear.
5. Voluntarily participate in the study and sign the informed consent form.
6. Have normal mental status and cognitive function, and be able to cooperate with the research process.

Exclusion Criteria:

1. Diagnosis of Meniere's disease, conductive hearing loss or objective tinnitus.
2. History of epilepsy or stroke.
3. Diagnosis of acoustic neuroma.
4. Severe sensorineural hearing loss.
5. Surgically or traumatically implanted ferromagnetic foreign bodies, including but not limited to pacemakers, neurostimulators, prosthetic metal heart valves, aneurysm clips (non-titanium alloy), intraocular metal foreign bodies, cochlear implants, metal prostheses, metal joints, fixed steel plates or steel pins.
6. Patients with active metal foreign bodies (metal implants, dentures, contraceptive rings), insulin pumps, etc., who have been evaluated in detail and are at risk for rTMS treatment.
7. Patients taking vestibular sedatives, antipsychotics, anxiolytics, antiepileptics, and ototoxic drugs.
8. Patients with a recent history of alcohol or drug abuse
9. Bell's palsy
10. Acute ear infection within the last 1 month
11. Inability to cooperate or complete the study process
12. Participation in another clinical trial within the last month.
13. Have any condition that may affect compliance or safety
14. Any other condition that, in the opinion of the investigator, makes enrollment in the study inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 5 days from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).
Tinnitus Handicap Inventory (THI) | 12 days from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).
Tinnitus Handicap Inventory (THI) | 30 days from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 5 days from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Visual Analogue Scale (VAS) | 12 days from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Visual Analogue Scale (VAS) | 30 days from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Minimum Masking Level (MML) | 5 days from baseline
  The MML assessment quantifies the minimum sound intensity required to mask the perception of tinnitus.
Minimum Masking Level (MML) | 12 days from baseline
  The MML assessment quantifies the minimum sound intensity required to mask the perception of tinnitus.
Minimum Masking Level (MML) | 30 days from baseline
  The MML assessment quantifies the minimum sound intensity required to mask the perception of tinnitus.
Tinnitus Loudness Matching (LM) | 5 days from baseline
  Used to measure tinnitus loudness. The level of intensity of an external sound that the patient perceives as equivalent to their tinnitus is used as the LM measurement.
Tinnitus Loudness Matching (LM) | 12 days from baseline
  Used to measure tinnitus loudness. The level of intensity of an external sound that the patient perceives as equivalent to their tinnitus is used as the LM measurement.
Tinnitus Loudness Matching (LM) | 30 days from baseline
  Used to measure tinnitus loudness. The level of intensity of an external sound that the patient perceives as equivalent to their tinnitus is used as the LM measurement.
Duration and intensity of residual inhibition (RI) for tinnitus | 5 days from baseline
  Used to measure the duration and intensity of RI for tinnitus.
Duration and intensity of residual inhibition (RI) for tinnitus | 12 days from baseline
  Used to measure the duration and intensity of RI for tinnitus.
Duration and intensity of residual inhibition (RI) for tinnitus | 30 days from baseline
  Used to measure the duration and intensity of RI for tinnitus.
Self-rating Anxiety Scale (SAS) | 5 days from baseline
  The SAS is a concise, validated tool for assessing anxiety levels in research and clinical settings. It comprises 20 items rated on a 4-point scale, summing to a total score indicating anxiety severity.
Self-rating Anxiety Scale (SAS) | 12 days from baseline
  The SAS is a concise, validated tool for assessing anxiety levels in research and clinical settings. It comprises 20 items rated on a 4-point scale, summing to a total score indicating anxiety severity.
Self-rating Anxiety Scale (SAS) | 30 days from baseline
  The SAS is a concise, validated tool for assessing anxiety levels in research and clinical settings. It comprises 20 items rated on a 4-point scale, summing to a total score indicating anxiety severity.
Athens Insomnia Scale (AIS) | 5 days from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
Athens Insomnia Scale (AIS) | 12 days from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
Athens Insomnia Scale (AIS) | 30 days from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, PhD, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China